CLINICAL TRIAL: NCT02553148
Title: Estimating the Global Need for Palliative Care for Children: A Cross Sectional Analysis
Brief Title: Estimating the Global Need for Palliative Care for Children
Status: Completed | Type: Observational
Sponsor: International Children's Palliative Care Network (Other)
Collaborators: UNICEF (Other)
Responsible Party: Sponsor
Other Study IDs: 0001
Record Dates: First submitted 2015-08-19; First posted 2015-09-17 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Cancer; Congenital Anomalies; Cardiovascular Disease; HIV
Keywords: prevalence; epidemiology; palliative care; pediatric
MeSH Terms: conditions — Neoplasms; Congenital Abnormalities; Cardiovascular Diseases | interventions — Health Services Needs and Demand

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (23):
- Argentina: One of the 23 countries studied
  Interventions: Other: Need for children's palliative care
- Armenia: One of the 23 countries studied
  Interventions: Other: Need for children's palliative care
- Australia: One of the 23 countries studied
  Interventions: Other: Need for children's palliative care
- Brazil: One of the 23 countries studied
  Interventions: Other: Need for children's palliative care
- China: One of the 23 countries studied
  Interventions: Other: Need for children's palliative care
- Egypt: One of the 23 countries studied
  Interventions: Other: Need for children's palliative care
- Ethiopia: One of the 23 countries studied
  Interventions: Other: Need for children's palliative care
- Germany: One of the 23 countries studied
  Interventions: Other: Need for children's palliative care
- India: One of the 23 countries studied
  Interventions: Other: Need for children's palliative care
- Indonesia: One of the 23 countries studied
  Interventions: Other: Need for children's palliative care
- Jordan: One of the 23 countries studied
  Interventions: Other: Need for children's palliative care
- Kenya: One of the 23 countries studied
  Interventions: Other: Need for children's palliative care
- Kyrgyzstan: One of the 23 countries studied
  Interventions: Other: Need for children's palliative care
- Malaysia: One of the 23 countries studied
  Interventions: Other: Need for children's palliative care
- Malawi: One of the 23 countries studied
  Interventions: Other: Need for children's palliative care
- Mexico: One of the 23 countries studied
  Interventions: Other: Need for children's palliative care
- Russia: One of the 23 countries studied
  Interventions: Other: Need for children's palliative care
- Serbia: One of the 23 countries studied
  Interventions: Other: Need for children's palliative care
- South Africa: One of the 23 countries studied
  Interventions: Other: Need for children's palliative care
- Tajikistan: One of the 23 countries studied
  Interventions: Other: Need for children's palliative care
- United Kingdom: One of the 23 countries studied
  Interventions: Other: Need for children's palliative care
- United States: One of the 23 countries studied
  Interventions: Other: Need for children's palliative care
- Zimbabwe: One of the 23 countries studied
  Interventions: Other: Need for children's palliative care

INTERVENTIONS:
Other: Need for children's palliative care — Need for children's palliative care

SUMMARY:
A cross-sectional analysis of prevalence data from a stratified sample of 23 countries used to estimate the global need for palliative care for children aged 0-19 years. Prevalence data, from the Institute for Health Metrics and Evaluation, was for 12 major diagnostic groups needing children's palliative care according to WHO and UNICEF guidelines.

DETAILED DESCRIPTION:
There is growing awareness that there are major gaps in access to children's palliative care (CPC) worldwide. Adults have a greater likelihood of receiving palliative care than children. Growing access to treatment services, and extended periods of wellness have led to some changes in the nature of the palliative care services required. Children are more resilient and more likely to require CPC for longer periods than adults.

It is against this background that UNICEF and the International Children's Palliative Care Network (ICPCN), in collaboration with national palliative care associations, began a joint analysis to develop methods to assess critical needs and gaps in CPC. The initial assessment, conducted in Kenya, South Africa and Zimbabwe, aimed to analyse existing secondary data on palliative care to estimate the palliative care need amongst children and explore key gaps in the response with service providers. A report on this research, the methods used, and the results for South Africa was published in 2014.

There is a lack of information regarding the actual need for palliative care for children, and assessment is a complicated process, due to uncertainty about the patient population and the nature of palliative care for children. Although there have been some studies focusing on the status of CPC in sub-Saharan Africa and the United Kingdom, there are differences in the scope and approach to the present study. A systematic review of the provision of CPC around the world, noted that over 65% of countries have no recognised CPC service provision, and concluded that service provision for CPC is not meeting the need in the majority of the world.

Generally, studies estimating need for palliative care for children are based on mortality statistics for chronic, incurable illnesses. Estimates focused on end-of-life care, as in the Global Atlas of Palliative Care at the End of Life do not account for the children that need palliative care well before the last year of life and underestimate the need.

The World Health Organization defines palliative care for children as a special, albeit closely related field to adult palliative care. An effort to define the many diseases and conditions requiring CPC a directory was published in 2013 with 376 potential diagnostic labels though the majority of deaths were from a small number.

ELIGIBILITY:
Inclusion Criteria:

* have one of the conditions above

Exclusion Criteria:

* greater than 19 years of age

Max Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: All children in sample countries with the following diagnoses included: all cancers (except non-malignant skin); HIV/AIDS; cardiovascular diseases; cirrhosis of liver; congenital anomalies; endocrine, blood, & immune disorders; meningitis; kidney diseases; protein energy malnutrition; neurological conditions; neonatal conditions; drug-resistant tuberculosis. Cases with sequela not associated with need for palliative care were removed.
Sampling Method: Probability Sample
Enrollment: 18837613 (Actual)
Dates: Start 2014-06; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Need for Children's Palliative Care | 1 year
  Estimation of need in a stratified sample of countries to derive a global estimate

CONTACTS AND LOCATIONS:
Overall Officials: Joan Marston, MA, RN, Study Chair — International Children's Palliative Care Network; Stephen R Connor, PhD, Principal Investigator — International Children's Palliative Care Network
Locations (1):
- International Children's Palliative Care Network, Fairfax Station, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
A manuscript reporting results has been prepared and is being reviewed for journal publication.

REFERENCES:
- [Background] Institute of Medicine (US) Committee on Palliative and End-of-Life Care for Children and Their Families; Field MJ, Behrman RE, editors. When Children Die: Improving Palliative and End-of-Life Care for Children and Their Families. Washington (DC): National Academies Press (US); 2003. Available from http://www.ncbi.nlm.nih.gov/books/NBK220818/ PMID 25057608
- [Background] Harding R, Brits H, Penfold S. Paediatric antiretroviral therapy outcomes under HIV hospice care in South Africa. Int J Palliat Nurs. 2009 Mar;15(3):142-5. doi: 10.12968/ijpn.2009.15.3.41093. PMID 19537535
- [Background] Connor S, Sisimayi C, Downing J, King E, Lim Ah Ken P, Yates R, Marston J. Assessment of the need for palliative care for children in South Africa. Int J Palliat Nurs. 2014 Mar;20(3):130-4. doi: 10.12968/ijpn.2014.20.3.130. PMID 24675539
- [Background] Hain R, Heckford E, McCulloch R. Paediatric palliative medicine in the UK: past, present, future. Arch Dis Child. 2012 Apr;97(4):381-4. doi: 10.1136/archdischild-2011-300432. Epub 2011 Oct 28. PMID 22039176
- [Background] Fraser LK, Miller M, Hain R, Norman P, Aldridge J, McKinney PA, Parslow RC. Rising national prevalence of life-limiting conditions in children in England. Pediatrics. 2012 Apr;129(4):e923-9. doi: 10.1542/peds.2011-2846. Epub 2012 Mar 12. PMID 22412035
- [Background] Knapp C, Woodworth L, Wright M, Downing J, Drake R, Fowler-Kerry S, Hain R, Marston J. Pediatric palliative care provision around the world: a systematic review. Pediatr Blood Cancer. 2011 Sep;57(3):361-8. doi: 10.1002/pbc.23100. Epub 2011 Mar 17. PMID 21416582
- [Background] Hain R, Devins M, Hastings R, Noyes J. Paediatric palliative care: development and pilot study of a 'Directory' of life-limiting conditions. BMC Palliat Care. 2013 Dec 11;12(1):43. doi: 10.1186/1472-684X-12-43. PMID 24330676